CLINICAL TRIAL: NCT00376207
Title: Physical Activity After Stroke: How Does it Effect Chronical Inflammation and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: LK-0102200601
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Cerebral Infarction
Keywords: Cerebral infarct; physical exercise; insulin sensitivity; low grade chronic inflammation; intervention; HOMA; PASE
MeSH Terms: conditions — Cerebral Infarction; Motor Activity; Insulin Resistance | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical exercise

SUMMARY:
Decreased insulin sensitivity is and independent risk factor for stroke despite glycemic control. It is known that physical exercise increases insulin sensitivity in healthy subjects. Wether stroke patients can increase insulin sensitivity via physical exercise is not known.

Chronic low-grade inflammation is associated with an increased risk of stroke. Physical exercise has shown to increase IL-6 directly after exercise in untrained subjects. When fitness is increased in each subject then the peak IL-6 concentration after exercise decreases and so does the basal level of IL-6. It is not known whether stroke patients can increase physical activity level to a degree where chronic inflammation are decreased.

This study is designed to evaluate if physical exercise after stroke will increases insulin sensitivity and reduce low-grade chronic inflammation.

Stroke patients have been randomized to intervention with physical exercise or control in the ExStroke pilot trial and followed for 2 years. Using the study population from the ExStroke pilot trail blood samples will be obtained at the last control. Insulin sensitivity can be measured from fasting glucose and insulin using the Homeostasis Model Assessment (HOMA). Interleukin-6, TNF-alfa and CRP is measured to estimate chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* participated in the ExStroke Pilot trail

Exclusion Criteria:

* Diabetes Mellitus
* Not able to give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Association between PASE and HOMA
Association between PASE and IL-6

SECONDARY OUTCOMES:
IL-6 concentration is lower in the intervention group than control group.
TNF-alfa and IL-6 is positively associated.
IL-18 is associated to HOMA
Correlation between PASE and HOMA in the intervention group vs. controls
HOMA mean value in the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Henrik Krarup, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark